CLINICAL TRIAL: NCT03773965
Title: A Phase 3 Multicenter Study to Evaluate the Long-Term Safety and Efficacy of Baricitinib in Patients From 1 Year to <18 Years of Age With Juvenile Idiopathic Arthritis (JIA)
Brief Title: A Study of Baricitinib in Participants From 1 Year to Less Than 18 Years Old With Juvenile Idiopathic Arthritis
Acronym: JUVE-X
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16278; I4V-MC-JAHX (Other: Eli Lilly and Company); 2017-004471-31 (EudraCT Number)
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Polyarticular JIA; Oligoarthritis; Juvenile psoriatic arthritis (JPsA); Enthesitis-related juvenile idiopathic arthritis (ERA); Systemic JIA with and without systemic features
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Baricitinib (Experimental): Baricitinib given orally.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104

SUMMARY:
The reason for this study is to see if the study drug baricitinib is safe and effective in the treatment of JIA in participants ages 1 to 17. This study is for participants that have been enrolled in studies I4V-MC-JAHV (NCT03773978) or I4V-MC-JAHU.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed a previous study of baricitinib for the treatment of JIA.

Exclusion Criteria:

* Participants must not have had a permanent discontinuation of baricitinib in the prior study.
* Participants must have not developed an allergy to baricitinib.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 190 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) | Baseline through Week 264
  Number of participants with one or more SAEs
Number of Participants with Permanent Investigational Product Discontinuations | Baseline through Week 264
  Number of participants with permanent investigational product discontinuations

SECONDARY OUTCOMES:
Proportion of Participants Achieving Pediatric American College of Rheumatology 30 Responder Index (PedACR30) | Week 264
  Proportion of participants achieving PedACR30
Proportion of Participants who have Disease Flare | Baseline through Week 264
  Proportion of participants who have disease flare
Proportion of Participants with Inactive Disease | Week 264
  Proportion of participants with inactive disease
Proportion of Participants with Minimal Disease Activity | Week 264
  Proportion of participants with minimal disease activity
Proportion of Participants in Remission | Week 264
  Proportion of participants in remission
Change from Baseline in Juvenile Arthritis Disease Activity Score-27 (JADAS27) | Baseline, Week 264
  Change from baseline of originating study in JADAS27
Change from Baseline in Arthritis-Related Pain Severity as Measured by the Childhood Health Assessment Questionnaire (CHAQ) Pain Visual Analog Scale (VAS) Item | Baseline, Week 264
  Change from baseline in arthritis-related pain severity as measured by the CHAQ pain VAS item
Change from Baseline in Psoriasis Area and Severity Index (PASI) | Baseline, Week 264
  Change from baseline in PASI
Change from Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index | Baseline, Week 264
  Change from baseline in SPARCC enthesitis index
Change from Baseline in Juvenile Spondyloarthritis Disease Activity Index (JSpADA) | Baseline, Week 264
  Change from baseline in JSpADA
Change from Baseline in Immunoglobulin Levels | Baseline, Week 264
  Change from baseline in immunoglobulin levels
Change from Baseline in Immunophenotyping (T Cells) | Baseline, Week 264
  Change from baseline in immunophenotyping (T Cells)
Change of Immunoglobulin G (IgG) Titers | Pre-Vaccination to 12 Weeks Post-Vaccination
  Change of IgG titers

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (82):
- Argentina (2):
  - Instituto CAICI SRL, Rosario
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman
- Australia (3):
  - Royal Children's Hospital, Melbourne
  - Perth Children's Hospital, Perth
  - The Children's Hospital at Westmead, Westmead
- Landeskrankenhaus Bregenz, Bregenz, Austria
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (5):
  - Faculdade de Medicina da UNESP, Botucatu
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - IPITEC, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo
  - Instituto da Crianca do Hospital das Clinicas da FMUSP, São Paulo
- China (4):
  - Beijing Children's hospital, Capital Medical University, Beijing
  - The Children's Hospital of Chongqing Medical University, Chongqing
  - Childrens Hospital of Nanjing Medical University, Nanjing
  - Children's Hospital of Soochow University, Suzhou
- Czechia (3):
  - Detska nemocnice FN Brno, Brno
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice Motol, Prague
- Aarhus Universitetshospital, Skejby, Aarhus, Denmark
- France (5):
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Bron
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
- Germany (6):
  - Helios Klinikum Berlin-Buch, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Praxis Kinder- und Jugendrheumatologie Dr. Ivan Foeldvari, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Asklepios Klinik Sankt Augustin, Sankt Augustin
  - Universitaetsklinikum Tuebingen, Tübingen
- India (3):
  - Sri Ramachandra MedicaL College & Research Institute, Chennai
  - Sir Ganga Ram Hospital, New Delhi
  - Christian Medical College Vellore, Vellore
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (8):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti, Chieti
  - IRCCS Istituto Giannina Gaslini, Genova
  - Centro Specialistico Ortopedico Traumatologico Gaetano Pini - CTO, Milan
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - University of Naples Federico II, Napoli
  - Azienda di Rilievo Nazionale e Alta Specializzazione Civico Di Cristina Benfratelli, Palermo
  - Ospedale Infantile Burlo Garofolo, Trieste
- Japan (11):
  - Institute of Science Tokyo Hospital, Bunkyō
  - Chiba Children's Hospital, Chiba
  - Kagoshima University Hospital, Kagoshima
  - Kanazawa University Hospital, Kanazawa
  - Niigata University Medical & Dental Hospital, Niigata
  - Saitama Children's Medical Center, Saitama-shi
  - Miyagi Children's Hospital, Sendai
  - Tokyo Women's Medical University Hospital, Shinjuku-ku
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Kanagawa Children's Medical Center, Yokohama
  - Yokohama City University Hospital, Yokohama
- Mexico (5):
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
  - Instituto de Investigaciones Clínicas para la Salud, Durango
  - Crea de Guadalajara, Guadalajara
  - Clinstile, S.A. de C.V., México
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey
- Poland (3):
  - Wojewódzki Specjalistyczny Szpital Dziecięcy im. św. Ludwika w Krakowie, Krakow
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji, Warsaw
- Russia (2):
  - Federal State Budgetary Scientific Institution Research Institute Rheumatology named after V.A.Nasonova, Moscow
  - Scientific Center of Children's Health, Moscow
- Spain (6):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpasa, Cerrahpasa Faculty of Medicine, Istanbul
  - 9 Eylul University Hospital, Izmir
- United Kingdom (5):
  - Bristol Royal Hospital for Children, Bristol
  - Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London
  - Oxford University Hospitals - Nuffield Orthopaedic Centre, Oxford
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Study of Baricitinib in Participants From 1 Year to Less Than 18 Years Old With Juvenile Idiopathic Arthritis — https://trials.lillytrialguide.com/en-US/trial/1jKB0Gb6daw6sUu4gseGga